CLINICAL TRIAL: NCT00602862
Title: The Effect of Sorafenib (Nexavar®) on 111-Indium Labeled Chimeric Monoclonal Antibody G250 or 111-Indium Labeled Bevacizumab (Avastin®) Uptake in Patients With Clear Cell RCC (ccRCC)
Brief Title: Effect of Sorafenib on ccRCC Uptake of Radiolabeled Bevacizumab or cG250
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Dutch Cancer Society (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Sorafenib-mAbs
Record Dates: First submitted 2008-01-03; First posted 2008-01-28 (Estimated); Last update posted 2013-12-02 (Estimated); Status verified 2012-02

CONDITIONS: Clear Cell Renal Cell Carcinoma
Keywords: Angiogenesis inhibitors
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Sorafenib; Bevacizumab; G250 monoclonal antibody; Indium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): 10 Patients planned to undergo (partial) nephrectomy or metastasectomy receive an iv injection of 100 MBq/1mg 111In-Bevacizumab. Patients are then treated with Sorafenib 200 mg 2dd2 po for 4 weeks. In the last week of treatment, the same injection is given to determine tumor accumulation of the radiolabeled mAb after Sorafenib treatment. Whole-body scintigraphic images are recorded 1 week after both injections to calculate tumor uptake. After Sorafenib treatment, patients will undergo surgery.
  Interventions: Drug: Sorafenib; Drug: 111Indium-bevacizumab
- 2 (Experimental): 10 Patients planned to undergo (partial) nephrectomy or metastasectomy receive an iv injection of 100 MBq/10mg 111In-cG250. Patients are then treated with Sorafenib 200 mg 2dd2 po for 4 weeks. In the last week of treatment, the same injection is given to determine tumor accumulation of the radiolabeled mAb after Sorafenib treatment. Whole-body scintigraphic images are recorded 1 week after both injections to calculate tumor uptake. After Sorafenib treatment, patients will undergo surgery.
  Interventions: Drug: Sorafenib; Drug: 111Indium-cG250
- 3 (Active Comparator): 5 Patients planned to undergo (partial) nephrectomy or metastasectomy receive an iv injection of 100 MBq/1mg 111In-Bevacizumab. Whole-body scintigraphic images are recorded 1 week after the injection to calculate tumor uptake. Hereafter, patients will undergo surgery.
  Interventions: Drug: 111Indium-bevacizumab

INTERVENTIONS:
Drug: Sorafenib — Sorafenib 200 mg 2dd2 po for 4 weeks before surgery
  Other Names: Bevacizumab; Avastin; Nexavar; cG250; Rencarex
  Arms: 1; 2
Drug: 111Indium-bevacizumab — 100 MBq / 1 mg 111Indium/bevacizumab iv
  Other Names: avastin; indium
  Arms: 1; 3
Drug: 111Indium-cG250 — 100 MBq / 10 mg 111Indium-cG250 iv
  Other Names: rencarex; indium
  Arms: 2

SUMMARY:
Sorafenib is a tyrosine kinase inhibitor that is registered for the treatment of metastasized clear cell Renal Cell Carcinoma (ccRCC). It inhibits signal transduction of the Vascular Endothelial Growth Factor Receptor (VEGFR) and the Platelet Derived Growth Factor Receptor (PDGFR). In the tumorigenesis of ccRCC, VEGF and PDGF are upregulated due to the defective Von-Hippel-Lindau (VHL) gene. CcRCC has a high Interstitial Fluid Pressure (IFP) and Tumor Microvascular Density (TMD), hampering the delivery of chemotherapeutics and monoclonal antibodies (mAbs). It was hypothesized that antiangiogenic compounds decrease tumor IFP and TMD, thus normalizing tumor vasculature, before diminishing tumor vasculature. Bevacizumab is an anti-VEGF mAb which depletes soluble VEGF from plasma, depriving VEGFR of its ligand. Chimeric monoclonal antibody cG250 recognizes carbonic anhydrase IX (CAIX), an antigen that is abundantly expressed in Renal Cell Carcinoma (RCC) and has limited expression in normal tissue. The aim of this study was to investigate the effect of Sorafenib on ccRCC physiology, by determining tumor uptake of 111In labeled cG250 or 111In labeled Bevacizumab.

ELIGIBILITY:
Inclusion Criteria:

* Renal cell carcinoma patients planned for surgery (nephrectomy/metastasectomy)
* Karnofsky > 70 %
* Laboratory values within 14 days prior to start:

  * White blood cells (WBC) > 3.5 x 109/L
  * Platelets > 100 x 109/L
  * Hemoglobin > 6 mmol/L
  * Total bilirubin < 1.5 upper limit of normal (ULN)
  * ASAT, ALAT < 2.5 x ULN (<5 x in case of liver metastases)
  * Lactate dehydrogenase (LDH) > 1.5. ULN
  * Serum creatinine < 2 x ULN
  * Amylase and Lipase < 1.5 ULN
* Negative pregnancy test in premenopausal women
* Age over 18 years
* Signed informed consent
* Life expectancy > 24 weeks
* PT/APTT/ INR < 1.5 ULN
* No current use of coumarin derivatives

Exclusion Criteria:

* Known subtype other than clear cell RCC
* Pre-exposure to murine/chimeric antibody therapy
* Known brain metastases
* Untreated hypercalcemia
* Uncontrolled hypertension
* Concurrent therapeutic anticoagulation
* Chemotherapy, immunotherapy or radiation therapy within 4 weeks prior to start of study. Palliative limited field external radiation for fracture prevention is allowed
* Cardiac arrhythmias requiring antiarrhythmics (beta-blockers, digoxin), symptomatic coronary artery disease and congestive heart failure New York Heart Association III or IV.
* Previous malignancy < 2 years prior to the study (except for cervical carcinoma in situ, basal cell carcinoma, or superficial bladder tumours (Ta, Tis, T1)
* Any medical condition present that in the opinion of the investigator will affect patients' clinical status. No other concurrent malignancy except nonmetastatic nonmelanoma skin cancer or carcinoma in situ of the cervix.
* Active clinically serious bacterial or fungal infections (< grade 2 NCI-CTC version 3)
* Known history of Human Immunodeficiency virus (HIV) infection or chronic hepatitis B/C.
* Prior use of Raf-kinase inhibitors, MEK and Farnesyl transferase inhibitors
* Prior use of Bevacizumab and all other drugs that target VEGF/ VEGF-receptors
* Use of antiepileptic drugs
* Pregnancy and lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2007-07; Primary Completion 2012-04 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
To determine the effect of sorafenib treatment on 111In-cG250 uptake of the tumor | pre-surgery
To determine the effect of sorafenib treatment on 111In-bevacizumab uptake of the tumor | pre-surgery

SECONDARY OUTCOMES:
Immunohistochemical analysis of CA-IX expression, (p)VHL status, HIF1-a, VEGF and PDGF expression, apoptosis and necrosis of surgical specimen | within 6 months post-surgery

CONTACTS AND LOCATIONS:
Overall Officials: WJG Oyen, MD, PhD, Principal Investigator — Department of Nuclear Medicine, Radboud University Nijmegen Medical Center, Nijmegen, The Netherlands; PFA Mulders, MD, PhD, Principal Investigator — Department of Urology, Radboud University Nijmegen Medical Center, Nijmegen, The Netherlands
Locations (1):
- Radboud University Nijmegen Medical Center, Nijmegen, Gelderland, Netherlands

REFERENCES:
- [Derived] Desar IM, Stillebroer AB, Oosterwijk E, Leenders WP, van Herpen CM, van der Graaf WT, Boerman OC, Mulders PF, Oyen WJ. 111In-bevacizumab imaging of renal cell cancer and evaluation of neoadjuvant treatment with the vascular endothelial growth factor receptor inhibitor sorafenib. J Nucl Med. 2010 Nov;51(11):1707-15. doi: 10.2967/jnumed.110.078030. Epub 2010 Oct 18. PMID 20956472